CLINICAL TRIAL: NCT03555903
Title: Quality of Life and Fertility of Patient With Deep Surgical Endometriosis: a Prospective Cohort
Acronym: ENDORAA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0813
Record Dates: First submitted 2018-01-23; First posted 2018-06-14 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Deep Infiltrating Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometriosis cohort: The aim of the study is to advance the scientific knowledge of deep infiltrating endometriosis (DIE) and to evaluate the impact of surgery on the quality of life and the fertility of affected women.
  Interventions: Other: Endometriosis cohort

INTERVENTIONS:
Other: Endometriosis cohort — The investigator record data on risks factors, symptoms (pain), quality of life (using standardized quality of life questionnaires), infertility history, and management of the disease with a 5-years follow up.
  Different surgical procedures exist to treat DIE and are they are described in the database, to allow comparison.

SUMMARY:
Endometriosis is a common gynaecologic disease affecting 5 to 15% women of reproductive age and up to 40% of infertile women. It is characterized by the presence of active endometrial tissue outside the uterine cavity, potentially causing invalidating chronic pelvic pain and infertility. It is therefore crucial to limit the progression and/or recurrence of the disease, and to improve the quality of life of affected women.

Deep infiltrating endometriosis (DIE), an advanced form of the disease, is defined by the invasion of an anatomical structure and organ close to the uterus (i.e. uterosacral ligament, rectovaginal space, recto-sigmoidal colon or bladder), or by a peritoneal invasion greater than 5mm. The management of DIE is unfortunately not yet based on high-level evidence data; it mainly depends on the localization of the disease, the extend of the invasion and the severity of the symptoms. In the absence of clear guidelines based on empirical data, the choice between surgical or medical treatment remains difficult and controversial.

To improve optimal DIE management, the investigators aim to create a prospective database reporting on DIE surgically treated in a teaching hospital in Lyon/France (Centre hospitalier universitaire Lyon Sud)

Data on known risks factors, symptoms (pain), quality of life, infertility history and disease management will be obtained using self-questionnaires, clinic, paraclinic, surgical and histological records as follow.

1. Each patient will be asked to fill in electronics protected on-line forms: the first one before surgery, followed by three follow-up forms at 1, 2 and 5 years after surgery.
2. The surgeon will be asked to fill in two electronic protected on-line forms: the first one at the time of surgery and the second one during a post-operative consultation (one month after surgery).

The questionnaires used in this study are similar to those used for the Endometriosis database "CIRENDO" (explain briefly what it is), which will ultimately allow us to pool the data from the 2 databases.

This French prospective study will advance the scientific knowledge on DIE surgical treatment and, by helping evaluate the impact of the surgery on the quality of life and fertility of affected women, will guide future recommendations for an optimal management of this invalidating disease.

ELIGIBILITY:
Inclusion Criteria:

* surgically management for deep endometriosis

Exclusion Criteria:

* No surgical management necessary
* Isolated Adenomyosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surgically managed for deep endometriosis in Centre hospitalier Lyon sud, Lyon, France
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The impact of the management of deep endometriosis on the quality of life | 5 years
  Evolution of SF 36 quality of life scores.
The impact of the management of deep endometriosis on the quality of life | 5 years
  Evolution of EHP-30 quality of life scores.

SECONDARY OUTCOMES:
Describe endometriosis | 5 years
  Description of the study population : Socio-demographic data
Describe risk factors of the disease. | 5 years
  Postoperative complications (DINDO classification)
Describe diagnostic delay of the disease. | 5 years
  Description of diagnostic.
Describe diagnostic management of the disease. | 5 years
  Description of therapeutic management : Diagnostic loadings
Impact of the management of deep endometriosis on the use of assisted reproductive therapy. | 5 years
  Impact on fertility.
Describe risk factors of the disease. | 5 years
  Recurrence of endometriosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Lyon sud, Pierre-Bénite, France